CLINICAL TRIAL: NCT05438303
Title: A Phase 1, Multi-center, Open-label, 3-arm, Fixed Sequence Study to Assess the Effect of Co-administration of AZD9833 on the Pharmacokinetics of Midazolam (CYP3A4/5 Substrate), of Omeprazole (CYP2C19 Substrate), of Celecoxib (CYP2C9 Substrate) and of Dabigatran Etexilate (P-gp Transporter Substrate) in Healthy Postmenopausal Female Volunteers
Brief Title: Study to Assess the Effect of Co-Administration of AZD9833 on the Pharmacokinetics of Midazolam, of Omeprazole, of Celecoxib and of Dabigatran Etexilate in Healthy Postmenopausal Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D8532C00004
Record Dates: First submitted 2022-05-19; First posted 2022-06-29 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: Drug-Drug interaction; Midazolam; Omeprazole; Dabigatran etexilate; Celecoxib; Postmenopausal; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; Midazolam; Omeprazole; Dabigatran; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (midazolam and omeprazole) (Experimental): Participants will receive single oral doses of midazolam and omeprazole together (Day 1 of Treatment Periods 1 and 3) and repeated doses of AZD9833 (Days 1 to 5 of Treatment Period 2 and Day 1 of Treatment Period 3)
  Interventions: Drug: AZD9833; Drug: Midazolam; Drug: Omeprazole
- Arm B (Dabigatran etexilate) (Experimental): Participants will receive single oral doses of dabigatran etexilate (Day 1 of Treatment Periods 1 and 2) and single oral dose of AZD9833 (Day 1 of Treatment Period 2)
  Interventions: Drug: AZD9833; Drug: Dabigatran Etexilate
- Arm C (Celecoxib) (Experimental): Participants will receive single oral doses of celecoxib (Day 1 of Treatment Periods 1 and 3) and repeated oral doses of AZD9833 (Days 1 to 5 of Treatment Period 2 and Day 1 of Treatment Period 3)
  Interventions: Drug: AZD9833; Drug: Celecoxib

INTERVENTIONS:
Drug: AZD9833 — AZD9833 tablets will be administered orally once daily on Days 1 - Day 5 (Treatment Period 2) and Day 1 (Treatment Period 3) for participants recruited to Arms A and C and Day 1 for those in Arm B
Drug: Midazolam — Midazolam will be administered orally as a syrup once on Day 1 of Treatment Periods 1 and 3; administered together with Omeprazole
  Arms: Arm A (midazolam and omeprazole)
Drug: Omeprazole — An Omeprazole capsule will be administered once on Day 1 of Treatment Periods 1 and 3; administered together with Midazolam
  Arms: Arm A (midazolam and omeprazole)
Drug: Dabigatran Etexilate — A Dabigatran Etexilate capsule will be administered once on Day 1 of Treatment Periods 1 and 2
  Arms: Arm B (Dabigatran etexilate)
Drug: Celecoxib — A Celecoxib capsule will be administered once on Day 1 of Treatment Periods 1 and 3
  Arms: Arm C (Celecoxib)

SUMMARY:
This study will be a fixed sequence drug-drug interaction study in healthy postmenopausal females, conducted at multiple study sites

DETAILED DESCRIPTION:
Participants will be randomized to one of 3 treatment arms on Day 1 prior to Investigational Medicinal Product (IMP) administration:

* Arm A: single oral doses of midazolam and omeprazole administered together + repeated doses of AZD9833 .
* Arm B: single oral doses of dabigatran etexilate + single oral dose of AZD9833 .
* Arm C: single oral doses of celecoxib + repeated oral doses of AZD9833.

Each participant will be involved in the study for up to 7 to 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal female participants aged 50 to 70 years with suitable veins for cannulation or repeated venipuncture.
* Participants must be postmenopausal by fulfilling the following criterion:
* Have a Body mass index (BMI) between 19 and 35 kg/m^2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive as measured at screening.
* Must agree to not use warfarin or phenytoin (and other coumarin-derived vitamin K antagonist anticoagulants) during study, and for 2 weeks after last administration of IMP.

Exclusion Criteria:

* History of any clinically significant disease or disorder as described by the Investigator.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Use of systemic estrogen-containing hormone replacement therapy within 6 months prior to first dose in the study.
* Have taken any proton pump inhibitors (omeprazole, lansoprazole, esomeprazole, pantoprazole, etc.) within 14 days of beginning study treatment (ie, first administration of omeprazole in Arm A.
* Have taken any drug with enzyme-inducing properties such as St John's Wort within 3 weeks of screening.
* Presence of any contraindication to the probe substrates omeprazole, midazolam, dabigatran or celecoxib per the United States Package Insert.
* Any of the following signs or confirmation of COVID-19 infection:
* Subject has a positive RT-PCR test for SARS-CoV-2 prior to randomization.
* Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnea, sore throat, fatigue) or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or at randomization.
* Subject has been previously hospitalized with COVID-19 infection within the last 12 months.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) of midazolam, omeprazole, total dabigatran, and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  The effects of AZD9833 will be evaluated in healthy postmenopausal female participants on the key pharmacokinetic (PK) variables of: - single-dose midazolam and omeprazole, administered together
  * single-dose dabigatran etexilate
  * single-dose celecoxib
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) of midazolam, omeprazole, total dabigatran, and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  The effects of AZD9833 will be evaluated in healthy postmenopausal female participants on the key pharmacokinetic variables of:
  * single-dose midazolam and omeprazole, administered together
  * single-dose dabigatran etexilate
  * single-dose celecoxib
Maximum observed plasma concentration (Cmax) of midazolam, omeprazole, dabigatran etexilate and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  The effects of AZD9833 will be evaluated in healthy postmenopausal female participants on the key pharmacokinetic variables of:
  * single-dose midazolam and omeprazole administered together
  * single-dose dabigatran etexilate
  * single-dose celecoxib

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From Screening until Post study (5 to 7 days post final dose) (assessed up to 6 months)
  The safety and tolerability of AZD9833, alone and in combination with midazolam, omeprazole, dabigatran etexilate, and celecoxib will be evaluated in healthy postmenopausal female participants.
AUCinf for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of dabigatran etexilate will be further characterized.
AUClast for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of dabigatran etexilate, and will be further characterized.
Area under plasma concentration-time curve in the dose interval (AUCt) for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of dabigatran etexilate will be further characterized.
Cmax for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of dabigatran etexilate will be further characterized
Time to reach maximum observed concentration (tmax) for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
Half-life associated with terminal slope of a semi-logarithmic concentration-time curve (t½λz) for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
Apparent total body clearance from plasma after extravascular administration (CL/F) for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
Apparent volume of distribution based on terminal phase (Vz/F) for AZD9833 and free dabigatran | For AZD9833 in Arm A: Day 1 and Day 2 (Period 3); For AZD9833 in Arm B: Day 1 and Day 2 (Period 2); For dabigatran: Day 1 to Day 3 (Period 1 and 2) (Each Period lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
tmax for midazolam, omeprazole, total dabigatran, and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
t½λz for midazolam, omeprazole, total dabigatran, and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
CL/F for midazolam, omeprazole, total dabigatran, and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
Vz/F for midazolam, omeprazole, total dabigatran, and celecoxib | For Arm A: Day 1 to Day 2 (Period 1 and 3); For Arm B: Day 1 to Day 3 (Period 1 and 2) (Each Period is 4 days); For Arm C: Day 1 to Day 4 (Period 1 and 3) (For Arm A and C, Period 1 is for 5 days and Period 3 is for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.
Area under the plasma concentration-curve from zero to 24 hours post dose (AUC0-24) for celecoxib | Day 1 to Day 4 (Period 1) (Period 1 lasts for 5 days) and Day 1 to Day 4 (Period 3) (Period 3 lasts for 4 days)
  AZD9833 PK and the effect of AZD9833 on the PK of midazolam, omeprazole, dabigatran etexilate, and celecoxib will be further characterized.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Long Beach, California
  - Research Site, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home